CLINICAL TRIAL: NCT07066605
Title: The Effect of Dexmedetomidine on Agitation During Weaning From Mechanical Ventilation in Critically Ill Patients"
Brief Title: The Effect of Dexmedetomidine on Agitation During Weaning From Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dalia Ayman Hussien, Resident, Department of Anesthesia, Intensive Care and Pain management, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-25-6---17MS
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dexmedetomidine
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Dexmedetomidine Group) (Active Comparator): patients will receive dexmedetomidine infusion starting at 0.2 mcg/kg/hr.
  Interventions: Drug: Group A (Dexmedetomidine Group)
- Group B (Control Group) (Placebo Comparator): patients will receive standard ICU sedation protocol without dexmedetomidine (e.g., fentanyl)
  Interventions: Drug: Group B (Control Group)

INTERVENTIONS:
Drug: Group A (Dexmedetomidine Group) — patients will receive dexmedetomidine infusion starting at 0.2 mcg/kg/hr.
  Arms: Group A (Dexmedetomidine Group)
Drug: Group B (Control Group) — patients will receive standard ICU sedation protocol without dexmedetomidine (e.g., fentanyl)
  Arms: Group B (Control Group)

SUMMARY:
This study aims to evaluate the effect of dexmedetomidine on the level of agitation during the weaning process from mechanical ventilation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients (≥18 years).
* On mechanical ventilation ≥24 hours.
* Clinically ready for weaning.
* Agitation score RASS ≥ +1 during spontaneous breathing trial.
* Intubation for at least 4 days: 2 weeks.

Exclusion Criteria:

* Known hypersensitivity to dexmedetomidine.
* Hemodynamic instability (HR < 50 bpm or MAP < 60 mmHg).
* Neurological impairment affecting level of consciousness.
* Pregnancy or lactation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Dexmedetomidine on Agitation During Weaning from Mechanical Ventilation | every half an hour for two hours
  Richmond Agitation-Sedation Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343